CLINICAL TRIAL: NCT01639352
Title: Phase II Trial of SOM230 (Pasireotide LAR) in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Phase II Trial of SOM230 in Patients With Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynn Feun (Other)
Responsible Party: Sponsor-Investigator, Lynn Feun, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100650
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; HCC; SOM230; Pasireotide LAR
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOM230 (Experimental): 60mg of SOM230 via injection intramuscularly every 28 days
  Interventions: Biological: SOM230

INTERVENTIONS:
Biological: SOM230 — Patients will be given a starting of 60mg of SOM230 via injection, intramuscularly every 28 days.
  Other Names: Pasireotide LAR; SOM230C

SUMMARY:
The hypothesis of this clinical trial is that hepatocellular carcinomas contain somatostatin receptors which make them sensitive to the inhibitory effects of a new somatostatin analog, SOM230. This analog has greater and broader binding affinity to somatostatin receptors compared to the current drug in use, sandostatin LAR. Thus, SOM230 has the potential to be more effective in the treatment of patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
For all patients, SOM230 will be given at a starting dose of 60 mg intramuscularly (IM) every 28 days. Dose reduction will be allowed for toxicities which are deemed to be therapy-related. Patients will receive SOM230C (IM) as an outpatient and will be observed for at least 30 minutes for any immediate adverse reactions. Toxicity checks will be done every 2 weeks and laboratory tests every 4 weeks during study therapy). Safety and efficacy will be assessed throughout the treatment period. Toxicities will be graded using the Common Terminology Criteria for Adverse Events, version 4.02.

Therapy will continue for maximum of two years if the patient shows no evidence of disease progression or intolerable toxicity. After completion of all study related therapy patients will complete a 30 day safety follow up visit. Patients who are still benefiting from therapy after two years may continue longer only after discussion between the Principal Investigator (PI) and the drug sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of unresectable HCC by either:

   * Histopathology or
   * Elevated serum Alpha-fetoprotein (AFP) >400 ng/ml and findings on magnetic resonance imaging (MRI) or CT scans characteristic of a primary liver tumor.
   * Findings on MRI or CT scans characteristic of a primary liver tumor in patients with cirrhosis
   * Tumors at least 1 cm or greater
2. Age ≥ 18 years.
3. Minimum of four weeks since any major surgery, completion of radiation,or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy).
4. Patients may have progressed on sorafenib or refused or were intolerant of sorafenib. A maximum of 2 prior lines of systemic therapy (including chemotherapy or targeted therapy) will be allowed. Prior locoregional therapy such as surgery, radiofrequency ablation or transarterial chemoembolization are also allowed (these will not be counted as systemic therapy), provided that progression has been documented after these therapies, and at least 4 weeks have elapsed since the last therapy.
5. Karnofsky performance status (KPS) of 80 or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy 12 weeks or more.
7. Adequate bone marrow function as shown by: Absolute neutrophil count (ANC) ≥ 1.2 x 10^9/L, Platelets ≥ 50 x 10^9/L
8. Adequate liver function as shown by: serum bilirubin < 1.5x upper limit of normal (ULN) and serum transaminases activity ≤ 3 x ULN. Serum PT =< 16 seconds.
9. Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN.
10. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation (can start after one day of initiation of lipid lowering drug) of appropriate lipid lowering medication.
11. Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
12. Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.
13. Child's A and early Child's B (no more than 7 points on the Child Pugh Classification).
14. Measurable disease by CT scan with contrast. If evaluable disease or measurable disease has been previously treated, this must show signs of tumor progression by CT. Measurable disease and evaluable disease will be defined by the RECISTguidelines (see section 9.0).
15. Patients with cirrhosis either radiologically or pathology with findings either by CT scan or MRI characteristic of primary liver cancer are eligible.

Exclusion Criteria:

1. Prior octreotide therapy or any somatostatin analog.
2. Chronic treatment with systemic steroids or another immunosuppressive agent.
3. Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry (ie. within 1 week of signing the informed consent).
4. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
5. Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
6. Patients with uncontrolled diabetes mellitus (defined as HgA1c > 7% or =8% despite therapy) or a fasting plasma glucose > 1.5 ULN. Note: At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.
7. Patients with symptomatic cholelithiasis
8. Patients who have congestive heart failure (NYHA Class III or IV), unstable angina,sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment.
9. Patients who are at high risk for cardiac arrhythmias as defined by any of the following:

   * Baseline QTcF > 470 msec
   * History of syncope or family history of idiopathic sudden death or long QT syndrome
   * Sustained or clinically significant cardiac arrhythmias
   * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade atrioventricular block (AV) block
   * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by uncontrolled diabetes, or Parkinson's disease), HIV, uncontrolled hypothyroidism or cardiac failure
   * Concomitant medication(s) known to increase the QT interval (see Appendix II)
10. Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot).
11. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    * Severely impaired lung function
    * Any active (acute or chronic) or uncontrolled infection/ disorders.
    * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
12. Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of pasireotide). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
13. Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR formulations
14. History of noncompliance to medical regimens
15. Patients unwilling to or unable to comply with the protocol or unable to give informed consent.
16. Patients with baseline Alanine transaminase (ALT) or Aspartate transaminase (AST) > 3x ULN.
17. Patients with baseline serum bilirubin > 1.5 x ULN.
18. Prothrombin time (PT) > 16 seconds and/or partial thromboplastin time (PTT) > 1.5 x ULN
19. History of or current alcohol misuse/abuse within the past 12 months.
20. Known gallbladder or bile duct disease, acute or chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Feun, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOM230
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SOM230
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 65 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20
Prior Therapies [Count of Participants; unit: Participants] — The types of therapies study participants received for the study disease prior to study enrollment. Participants may have had multiple therapies.
  Participants
    No prior therapy | 2
    Transarterial chemoembolization (TACE) | 12
    Chemotherapy | 2
    Ablation | 6
    Ytrium 90 | 2
    Cryoablation | 1
    Sorafenib | 14
BCLC Staging [Count of Participants; unit: Participants] — Barcelona Clinic Liver Cancer (BCLC) staging classifies hepatocellular carcinoma (HCC) into five stages, based on the extent of study disease, Child-Pugh score, and ECOG performance status as follows:
  * Stage 0 (Very early stage)
  * Stage A (Early stage)
  * Stage B (Intermediate Stage)
  * Stage C (Advanced Stage)
  * Stage D (Terminal Stage)
  Participants
    BCLC Stage 0 | 0
    BCLC Stage A | 0
    BCLC Stage B | 5
    BCLC Stage C | 15
    BCLC Stage D | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: The disease-control rate (DCR) is defined as the proportion of participants achieving a best overall response of complete response (CR), partial response or stable disease (SD) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by MRI or CT Scan, and that is maintained for at least 8 weeks. CR is defined as disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; and SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: At least 2 cycles, about 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230
Number analyzed (Participants) | 20
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 9

2. Secondary Outcome: Rate of Progression-Free Survival (PFS):
Description: Rate of Progression-Free Survival (PFS). PFS will be measured from the date of enrollment to the earliest date of documented disease progression or death from any cause, whichever is earlier. Progression is defined according to RECIST v 1.1 criteria as an at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. For patients who remain alive without progression, follow up time will be censored at the date of last disease assessment.
Time Frame: From Enrollment Until Study Completion, Approximately 3 Years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SOM230
Number analyzed (Participants) | 20
months | 3 [2 to 4]

3. Secondary Outcome: Rate of Overall Survival (OS)
Description: Rate of Overall Survival (OS) in participants receiving protocol therapy. OS will be measured from the date of enrollment to the date of death or last contact.
Time Frame: From Enrollment Until Study Completion, Approximately 3 Years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SOM230
Number analyzed (Participants) | 20
months | 9 [4 to NA] — Seven patients were alive at the discontinuation of the study.

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Proportion of patients achieving Complete Response and Partial Response (CR+PR) to protocol therapy per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT Scan. CR is defined as disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230
Number analyzed (Participants) | 20
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0

5. Secondary Outcome: Duration of Overall Response
Description: Duration of Overall Response in participants achieving complete response (CR) or partial response (PR) to SOM230 treatment. The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Overall response is assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by MRI or CT Scan. CR is defined as disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Up to 2 Years
Population: No participants achieved complete response (CR) or partial response (PR) to protocol therapy.
Arm/Group | SOM230
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicity Profile of Protocol Therapy
Description: Number of patients experiencing adverse events and/or toxicities while receiving protocol therapy.
Time Frame: Up to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | SOM230
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: The period of adverse event collection will be from the day of the 1st treatment until at least 4 weeks after study discontinuation, up to 3 years.
Arm/Group | SOM230
All-Cause Mortality (participants affected / at risk) | 13/20
Serious Adverse Events (participants affected / at risk) | 5/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230 (N=20)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Obstruction, GI (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOM230 (N=20)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (5)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (6)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 4 (5)
Blood bilirubin increased (Investigations) | 2 (10)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Metabolism and nutrition disorders) | 1 (3)
Creatinine increased (Investigations) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 4 (4)
Edema: limb (Blood and lymphatic system disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 7 (8)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 2 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Aphthous Ulcer
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hemorrhage, GI (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (16)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Musculoskeletal and connective tissue disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 2 (2)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) — Lactic Acidosis
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 6 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1)
Scleral disorder (Eye disorders) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Ventricular Arrythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight Gain (Investigations) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes